CLINICAL TRIAL: NCT00090701
Title: A Phase 2, Open-Label, Multicenter Study Of The GARFT Inhibitor AG2037 In Patients With MetastatIC Non Small Cell Lung Cancer Who Failed Two Or Three Prior Treatments
Brief Title: A Phase 2, Open-Label, Multicenter Study of the GARFT Inhibitor in Patients With Metastatic Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4371005
Record Dates: First submitted 2004-09-02; First posted 2004-09-06 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

INTERVENTIONS:
Drug: AG2037

SUMMARY:
The primary objective of this study is to determine safety and activity of a novel anticancer agent in patients with metastatic non-small cell lung cancer who failed 2 or 3 prior systemic treatments.

ELIGIBILITY:
Inclusion Criteria:

* presence of measurable, metastatic non-small cell lung cancer (histologically or cytologically confirmed at the time of original diagnosis)
* treatment failure (recurrence, disease progression, or intolerable toxicity) of 2 or 3 prior systemic treatments. (Note: no more than 3 prior systemic regimens for non-small cell lung cancer including adjuvant chemotherapy)
* capable of understanding the nature of the trial and willing to give written informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* hemoglobin level of >=9 g/dL, absolute granulocyte count of >=1.5 × 109/L, and platelet count of >=100 × 109/L
* adequate renal function, as documented by a serum creatinine level of <=1.5 times the institutional upper limit of normal (ULN) and a measured or calculated creatinine clearance of >=60 mL/min
* adequate liver function, as demonstrated by a total bilirubin level of <=1.5 times ULN; levels of serum glutamate oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) <=2 times ULN. If the patient has liver involvement then AST and ALT should be <=5 times ULN
* for men with partners of child-bearing potential and all women of childbearing potential, willingness to use adequate contraception or practice abstinence during the course of the study at least 18 years of age
* life expectancy estimated at greater than 12 weeks

Exclusion Criteria:

* history of blood transfusion within the last 14 days
* need of concurrent administration of allopurinol
* history of radiotherapy or chemotherapy within 4 weeks (nitrosourea or mitomycin C within 6 weeks) of the anticipated first day of dosing (patient must be fully recovered from the acute effects of any prior chemotherapy or radiotherapy)
* any psychological or sociological condition, addictive disorder, or family problems that might preclude compliance with the protocol
* any unstable or severe intercurrent medical condition that in the opinion of the investigator might interfere with achievement of study objectives
* receipt of an investigational agent within 28 days before the anticipated first day of dosing (patient must have recovered from all acute effects of previously administered investigational agents)
* pregnant or breast-feeding
* previous treatment with GARFT inhibitors
* history of radiation therapy to more than 40% of the marrow space
* history of a malignancy (other than non-small cell lung cancer) except those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years
* active brain metastases (requiring treatment or progressing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-09

PRIMARY OUTCOMES:
To determine the overall objective response rate (complete and partial responses) of AG-2037 in patients with metastatic non-small cell lung cancer who failed 2 or 3 prior systematic treatments.

SECONDARY OUTCOMES:
Evaluate the safety of AG-2037.
Estimate the time to progression (TTP).
Evaluate 1-year overall survival of patients treated with AG-2037.
Evaluate population PK and correlate the various genetic markers of MTAP, folate, and purine metabolism with clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, New York, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4371005&StudyName=A+Phase+2%2C+Open%2DLabel%2C+Multicenter+Study+of+the+GARFT+Inhibitor+in+Patients+with+Metastatic+Non%2DSmall+Cell+Lung+Cancer